CLINICAL TRIAL: NCT04164576
Title: Study of the Pathogenicity and Humoral Immune Response Induced by BK Virus in Lung Transplant Recipients
Acronym: BKV-Pneumo
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7547
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Renal-urinary Impairment; Graft Rejection; Infection Episodes
Keywords: Lung transplantation; BKV; Nephropathy; Immunosuppression
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum, white cells, urine, bronchoalveolar fluid, frozen and fixed tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Transplant patients — Study the specific immunity against Polyomavirus

SUMMARY:
BK virus (BKV) is a ubiquitous virus that infects more than 80% of the population. In case of immunosuppression, BKV can replicate and induce nephropathies in renal transplant recipients or haemorrhagic cystitis in bone marrow transplant recipients. The disruption of the balance between BKV replication and immune control is considered the key element in the development of these pathologies. During lung transplantation, patients undergo intense immunosuppression that favors the reactivation of persistent viruses such as EBV, CMV and probably BKV. Although the data on EBV and CMV reactivation are very clear and allow optimal management, the prevalence of BKV replication and its clinical impact in lung transplant recipients remains unknown at this time.

The aim of this study is to know the incidence and clinical impact of BKV replication in lung transplant recipients. Moreover, the results will help to better understand the interaction between the virus and his host, with a focus on the humoral and cellular immune response against BKV. The results could possibly enable to define predictive markers of BKV replication and of its evolution.

ELIGIBILITY:
Inclusion criteria:

* Lung transplant recipients in Strasbourg University Hospital between 30 June 2018 and 31 December 2022
* Male or female patients, age over 18 years
* Patient having provided informed written consent to take part in the study
* Patient affiliated to Social Security

Exclusion criteria:

* Patient deprived of liberty, by judicial or administrative decision
* Patient under legal guardianship
* Impossibility to give complete information about this study to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients between 30 June 2018 and 31 December 2022 at the University Hospital of Strasbourg
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
BKV viral load in urine (viruria) and in plasma (viremia) | 3 years
  In cases of positive viral load, the viral genome will be sequenced to identify the replicative genotype.

SECONDARY OUTCOMES:
Quantification of anti-BKV neutralizing antibodies | 3 years

OTHER OUTCOMES:
Quantification of BKV specific T lymphocytes | 3 years
TTV viral load in plasma | 3 years
  Evaluation of the viral load of TTV (reflection of global immunosuppression) or its genotype (established by sequencing).

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided